CLINICAL TRIAL: NCT05585931
Title: Evaluate the Acute Effects of a Single Oral Dose of TPN171H on Semen Function in Healthy Male Subjects in China
Brief Title: Effect of TPN171H on Spermatogenesis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TPN171H-12
Record Dates: First submitted 2022-09-18; First posted 2022-10-19 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): 9 subjects receive 10 mg TPN171H for Period 1; Placebo for Period 2
  Interventions: Drug: TPN171H 10mg; Drug: TPN171H Placebo
- Cohort 2 (Experimental): 9 subjects receive Placebo for Period 1; 10 mg TPN171H for Period 2
  Interventions: Drug: TPN171H 10mg; Drug: TPN171H Placebo

INTERVENTIONS:
Drug: TPN171H 10mg — Subjects were given 10mg TPN171H tablet with 240 mL warm water under fasting condition.
Drug: TPN171H Placebo — Subjects were given Placebo with 240 mL warm water under fasting condition.

SUMMARY:
This study is a phaseⅠstudy to determine the acute effects of TPN171H on semen function in healthy male subjects.

DETAILED DESCRIPTION:
Safety Study in male subjects

ELIGIBILITY:
Inclusion Criteria:

1. Male aged 18~40years (included)
2. Body Mass Index of 19 to 28 kg/m2; Body weight no less than 50 kg;
3. Sperm concentration ≥15*10^6/ml, Sperm motility(a+b(%))≥32%, Semen volume ≥1.5 ml, Liquefaction time≤60 min
4. Sperm sample should be collected after a minimum of 2 days and a maximum of 7 days of sexual abstinence.
5. Take reliable contraceptive measures
6. Physical examination, vital signs examination, laboratory examination, ECG were normal or abnormal without clinical significance;
7. Be able to understand and willing to sign the Informed Consent Form;

Exclusion Criteria:

1. People with azoospermia, teratozoospermia, moderate-to-severe asthenozoospermia, and moderate-to-severe oligozoospermia and other abnormal semen disease
2. People with vasectomy and ligation
3. People who have a history of hypersensitivity to other PDE5 inhibitors or TPN171H;
4. There are clear diseases of the central nervous system, cardiovascular system, digestive system (including those with severe fatty liver in B-ultrasound examination), respiratory system, urinary system, blood system, metabolic disorders, etc. and require medical intervention or other unsuitable clinical trials Those with tested diseases (such as history of mental illness, etc.); those with a history of orthostatic hypotension;
5. Blurred vision or a history of the following ocular diseases: nonvascular anterior ischemic optic neuropathy (NAION), abnormal color vision, hereditary retinal degeneration (such as retinitis pigmentosa), macular degeneration;
6. A history of fainting needles or fainting blood;
7. Blood loss or blood donation of 400 mL or more within 3 months before administration;
8. Those who have taken any prescription drugs, over-the-counter drugs, Chinese herbal medicines or health care products within 2 weeks before administration
9. those who have participated in other drug clinical trials and received trial drugs within 3 months before
10. Positive results of alcohol breath test, or current/previous alcoholics (drinking more than 21 standard units per week. 1 standard unit contains 14 g of alcohol, such as 360 mL of beer or 45 mL of 40% spirits or 150 mL wine);
11. Urine drug screening positive；
12. Smoking more than 10 cigarettes per day ；
13. Those who are positive for hepatitis B surface antigen (HBsAg), HCV antibody, syphilis antibody and HIV antibody;
14. he investigator believes that there are other factors that are not suitable for participating in this trial.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Effect on semen function | 1.5 hours after taking the medicine
  The parameters of semen routine analysis were compared between TPN171H tablets and placebo.
Seminal plasma exposure | 1.5 hours after taking the medicine
  TPN171H exposure in seminal fluid

SECONDARY OUTCOMES:
Adverse events | From administration of study drug through 3 days after last administration of study drug
  adverse events (each study visit); laboratory evaluations; electrocardiogram and physical examination; vital signs will be assessed at various times during the study

CONTACTS AND LOCATIONS:
Overall Officials: Hui Jiang, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Yang Y, Zhang Z, Li L, Jiang Z, Juan J, Duan H, Wang Z, Jiang H. Evaluation of the acute effects of single-dose TPN171 on semen quality in healthy Chinese male volunteers. Br J Clin Pharmacol. 2025 Aug;91(8):2401-2408. doi: 10.1002/bcp.70049. Epub 2025 Apr 3. PMID 40181588